CLINICAL TRIAL: NCT02582541
Title: Endoscopic Biliary Radiofrequency Ablation of Malignant Bile Duct Obstruction
Brief Title: Endoscopic Biliary RFA of Malignant Bile Duct Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFA-CN-1510
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Cholangiocarcinoma; Bile Duct Obstruction
MeSH Terms: conditions — Cholangiocarcinoma; Cholestasis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SEMS alone (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) was performed under standard operating conditions with a duodenoscope (TJF 260V, Olympus, Tokyo, Japan) to confirm the length of the biliary stricture, diameter, and position. An uncovered self expanding metallic stent (SEMS) (Wallstent, Boston Scientific, USA) would be placed across the biliary stricture.
  Interventions: Procedure: SEMS alone
- SEMS plus radiofrequency ablation (Experimental): Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the length of the biliary stricture, diameter, and position. The Habib EndoHBP catheter (Emcision, London, United Kingdom) was placed through the biliary stricture under fluoroscopic guidance. The RFA energy can be delivered repetitively at different tumor sites within one procedure, according to the stricture size. After the RFA application is completed, SEMS (Wallstent, Boston Scientific, USA) can be deployed.
  Interventions: Procedure: SEMS plus radiofrequency ablation

INTERVENTIONS:
Procedure: SEMS alone — The SEMS (Wallstent, Boston Scientific, USA) would be placed.
  Arms: SEMS alone
Procedure: SEMS plus radiofrequency ablation — The RFA catheter has an 8 F bipolar probe and two ring electrodes 8 mm apart with the distal electrode 5 mm from the leading edge, providing local coagulative necrosis over a 2.5 cm length. The catheter is compatible with standard side-viewing endoscopes (3.2 mm working channel), and could be passed over 0.035 inch guidewires. Ablation was performed by using an RFA generator (1500 RF generator; RITA Medical Systems, Fremont, Calif) delivering electrical energy at 400 kHz set at 7-10 W for 90-120 seconds. The RFA energy can be delivered repetitively at different tumor sites within one procedure. After the RFA application is completed, SEMS (Wallstent, Boston Scientific, USA) can be deployed.
  Arms: SEMS plus radiofrequency ablation

SUMMARY:
Endoscopic radiofrequency ablation (RFA) is a new palliation therapy for malignant bile duct obstruction. It delivers a high amount of thermal energy to target tissue and may prolong the duration of stent patency. RFA has showed promising results for malignant bile duct obstruction and increasing the duration of stent patency. The aim of our study was to evaluate the feasibility and safety of endoscopic RFA for the treatment of bile duct obstructions, and to compare the efficacy of Endoscopic biliary RFA with the addition of self-expanding metal stents (SEMS) to SEMS alone in a randomized controlled trial.

DETAILED DESCRIPTION:
Malignant bile duct obstructions are caused by many diseases arising from primary or metastatic disease in intrahepatic, extrahepatic or hilar locations. To relieve obstructive decompression and jaundice as a result of the obstruction, endoscopic stent placement is usually required. Compared with surgical intervention, stent insertion offers shorter hospitalization, lower overall cost and lower morbidity. Previous studies have shown the superiority of SEMSs over plastic stents for maintaining biliary drainage. However, SEMS can occlude due to epithelial hyperplasia, tumor in-/overgrowth, biofilm deposition and sludge formation. Studies have showed that the median SEMS patency is 120 days. Once bile duct obstruction reoccurs, it may lead to significant morbidity and mortality. Thus, long-term patency of the SEMS remains an unresolved issue.

Recently, endoscopic biliary radiofrequency ablation (RFA) have been used in patients suffering from inoperable malignant bile duct obstruction, and increasing the duration of stent patency. It delivers a high amount of thermal energy to target tissue with curative or palliative intent. The purpose of this study is to record information and evaluate the impact of radiofrequency ablation in improving the management of cholangiocarcinoma or malignant bile duct obstruction, and to compare the effects of SEMS plus RFA to SEMS alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically (preferred) or radiologically confirmed distal malignant bile duct tumors
2. Inoperability by staging, comorbidities or patient wishes

Exclusion Criteria:

1. History of bleeding disorder or use of anticoagulation
2. prior cardiac pacemaker placement
3. Presence of serious dysfunction of heart, lung or kidney.
4. Presence of other malignancy
5. Pregnancy
6. Prior SEMS placement
7. Prior Billroth II or roux-en Y reconstruction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Stent patency rate | 6 months

SECONDARY OUTCOMES:
Overall survival | 3 years
Number of Participants with Adverse Events | 30 days
Change from Baseline in Bile Duct Stricture Diameter | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Miao, MD, Principal Investigator — Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Wang F, Li Q, Ge X, Yu H, Nie J, Miao L. Choledochoscopic radiofrequency ablation for congenital choledochal cysts. Endoscopy. 2014;46 Suppl 1 UCTN:E373-4. doi: 10.1055/s-0034-1367604. Epub 2014 Sep 25. No abstract available. PMID 25254582
- [Background] Steel AW, Postgate AJ, Khorsandi S, Nicholls J, Jiao L, Vlavianos P, Habib N, Westaby D. Endoscopically applied radiofrequency ablation appears to be safe in the treatment of malignant biliary obstruction. Gastrointest Endosc. 2011 Jan;73(1):149-53. doi: 10.1016/j.gie.2010.09.031. PMID 21184881
- [Background] Wadsworth CA, Westaby D, Khan SA. Endoscopic radiofrequency ablation for cholangiocarcinoma. Curr Opin Gastroenterol. 2013 May;29(3):305-11. doi: 10.1097/MOG.0b013e32835faacc. PMID 23449026